CLINICAL TRIAL: NCT04592315
Title: A Study to Assess the Safety, Tolerability and Pharmacokinetics of Lipovirtide in HIV-infected Patients Without Prior Antiviral Therapy
Brief Title: A Study to Assess the Safety, Tolerability and Pharmacokinetics of Lipovirtide in HIV-infected Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanxi Kangbao Biological Product Co., Ltd. (Industry)
Collaborators: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KB-LP-80-101
Record Dates: First submitted 2020-09-30; First posted 2020-10-19 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-06

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- 1 (Experimental): Dose 5 mg
  Interventions: Drug: Lipovirtide Injection
- 2 (Experimental): Dose 10 mg
  Interventions: Drug: Lipovirtide Injection
- 3 (Experimental): Dose 20 mg
  Interventions: Drug: Lipovirtide Injection
- 4 (Experimental): Dose 40 mg
  Interventions: Drug: Lipovirtide Injection
- 5 (Experimental): Dose 60 mg
  Interventions: Drug: Lipovirtide Injection
- 6 (Experimental): Dose 80 mg
  Interventions: Drug: Lipovirtide Injection

INTERVENTIONS:
Drug: Lipovirtide Injection — Single dosage of Lipovirtide Injection

SUMMARY:
To evaluate the safety, tolerability of single dose lipovirtide injection in HIV-infected individuals without prior antiviral treatment, and to investigate the pharmacokinetic characteristics of infected patients.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged from 18 to 60 (include 18 and 60)；
2. Body mass index (BMI) [weight (kg)/ height 2(m2)] is from 18.0 to 26.0（include 18.0 and 26.0），male weight≥50kg，female weight≥45kg；
3. Confirmed HIV-1 infection；
4. HIV viral load ≥ 1000 copies/mL；
5. Patients who have no birth plan within 2 weeks before the screening and 3 months after the end of the trial, consenting to take effective non-drug contraceptive measures during the trial period；
6. Understand the purpose of and procedures required for the study and having confirmed they are willing to participate in the study by signing the informed consent document.

Exclusion Criteria:

1. Patients in the acute infection stage;
2. Confirmed AIDS patients；
3. Patients who have received antiviral therapy and/or have been vaccinated against HIV；
4. HBsAg is (+), and/or anti-HCV is (+)；
5. Abnormal liver function tests (ALT and / or AST> 3ULN, or total bilirubin> 2ULN)；
6. Glomerular filtration rate <70mL/min/1.73m2, or creatinine ≥ULN；
7. Patients who is currently suffering from a more serious chronic diseases, metabolic diseases (such as diabetes), neurological and mental diseases；
8. Patients who have previous history of pancreatitis；
9. Females who are pregnant or breastfeeding, or females of childbearing age who are unable to take contraception as required;
10. Allergic constitution or known allergy to the components of study drug；
11. With a history of smoking addiction within 12 months before screening (average number≥5 cigarettes per day)；
12. With a history of alcohol abuse within 12 months before screening (average drinking≥14 units of alcohol per week: 1 unit = 285mL beer, 25mL spirits, or 150mL wine) or those who have a positive alcohol breath test before enrollment；
13. With a history of drug abuse within 12 months before screening or those who tested positive for addictive substances before enrollment；
14. Patients who have participated in other investigational drug study within 3 months before screening (except for traditional Chinese medicine）；
15. Other factors that the investigators consider unsuitable for the trial.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2021-01-23 (Actual); Primary Completion 2023-05-02 (Actual); Study Completion 2023-07-11 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics：Cmax | Day 0 to Day 7
  pharmacokinetic characteristics of Lipovirtide in infected patients：Cmax
Pharmacokinetics：AUC0-t | Day 0 to Day 7
  pharmacokinetic characteristics of Lipovirtide in infected patients：AUC0-t

CONTACTS AND LOCATIONS:
Overall Officials: Haibin Yu, MD, Principal Investigator — Beijing You'an Hospital, Beijing Medical University; Hao Wu, MD, Principal Investigator — Beijing You'an Hospital, Beijing Medical University
Locations (1):
- Beijing You'an Hospital, Beijing Medical University, Beijing, Beijing Municipality, China